CLINICAL TRIAL: NCT04598139
Title: Safer Use of Medication in Pediatric Patients at Home: Error Reporting Website
Brief Title: Safer Use of Medication in Pediatric Patients at Home
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Mercedes Guilabert Mora, Principal investigator, Universidad Miguel Hernandez de Elche
Other Study IDs: PI18/00739
Record Dates: First submitted 2020-10-08; First posted 2020-10-22 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Medication Errors and Other Product Use Errors and Issues

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group
  Interventions: Other: Study group

INTERVENTIONS:
Other: Study group — The study group uses a web-based medication error notification system

SUMMARY:
This study aims:

* to develop a web-based notification system for caregivers of pediatric patients that allows to report medication errors and, based on this notification, and to share experiences and alerts about common errors of patients.
* to assess de user satisfaction and perceived usefulness of the system.

Participants:

Parents with children who have required drug treatment in the last two months, who have an Internet connection and who agree to participate in the study.

Sample size: 62 participants

Main outcome variable: overall satisfaction

ELIGIBILITY:
Inclusion Criteria:

* To care children aged under 14 years who have required drug treatment in the last two months
* To have an Internet connection
* To agree to participate in the study.
* To be registered in the study web-based notification system
* Age > 17 years

Exclusion Criteria:

* To be health provider
* To care children in residence for minors.
* To care children with a life expectancy of less than 2 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parents or caregivers of children aged from 0 to 14 years.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with the web-based medication error notification system | At one month after use of the website
  Overall satisfaction with the web-based medication error notification system by an ad hoc questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Mercedes Gilabert, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided